CLINICAL TRIAL: NCT02240901
Title: Effectiveness and Pulmonary Complications of Peri-Operative Laryngeal Mask Airway Used in Elderly Patients(POLMA-EP Trial): a Multi-center Randomized Controlled Clinical Trial
Brief Title: A Multi-center Randomized Clinical Trial About Using LMA or ETI in Elderly Patients
Acronym: LMA;ETI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Fudan University (Other); Shanghai Changzheng Hospital (Other); Shanghai First Maternity and Infant Hospital (Other); Huadong Hospital (Other); West China Hospital (Other); Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); Shanghai Jiading District Central Hospital (Other); Shanghai Pudong New Area Gongli Hospital (Other); Shanghai Huangpu District Central Hospital (Unknown); Shanghai Fengxian District Central Hospital (Other); People's Hospital of Pudong New District (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Wuxi No. 2 People's Hospital (Other); The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, LiqunYang, Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EHBH2013-003-005; EHBHKY20I3-003-005 (Other: EHBH)
Record Dates: First submitted 2014-08-23; First posted 2014-09-16 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: Complications; Surgery
Keywords: Laryngeal mask airway; endotracheal intubation; postoperative pulmonary complications; elderly patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Laryngeal mask airway (Experimental): Laryngeal mask airway（LMA） is used to maintain mechanical ventilation during intra-operative
  Interventions: Device: Laryngeal mask airway（LMA）
- Endotracheal intubation group（ETI） (Experimental): Endotracheal intubation group（ETI）is used to maintain mechanical ventilation during intra-operative
  Interventions: Device: Endotracheal intubation（ETI）

INTERVENTIONS:
Device: Laryngeal mask airway（LMA） — Laryngeal mask airway（LMA） is used to maintain mechanical ventilation during intra-operative
  Arms: Laryngeal mask airway
Device: Endotracheal intubation（ETI） — Endotracheal intubation group（ETI）is used to maintain mechanical ventilation during intra-operative
  Arms: Endotracheal intubation group（ETI）

SUMMARY:
Perioperative airway management is a top priority of anesthesiologists in daily work, and endotracheal intubation (ETI) is considered as the gold standard for providing safe glottic seal,effective ventilation and oxygen supplement during general anesthesia. But ETI related complications such as concomitant hemodynamic responses, damage to the oropharyngeal structures at insertion and postoperative sore throat. Laryngeal mask airway(LMA) for the anesthesia management brings new choice with invasive, lighter cardiovascular reaction and many other advantages, particularly suited to short and minimally invasive surgery. But LMA increased the risk of gastrointestinal reflux aspiration than using ETI and it may resulted in intolerance in high airway pressure, especially in elderly patients with increased lung compliance or reduced airway resistance. Furthermore, LMA could not entirely prevent the occurrence of postoperative sore throat and hoarse.

To sum up, it is necessary to carry out a multicenter clinical trial to clarify the safety of LMA in elderly patients. The investigators protocol will focus on the incidence of postoperative pulmonary complications (PPCs) when applications of LMA and ETI in elderly patients.

DETAILED DESCRIPTION:
1. Introduction 1.1 Background It is essential for peri-operative patients to ensure airway patency and effective ventilation, and respiratory is the most important task in anesthesiologist's daily work. Endotracheal intubation(ETI) is the gold standard for maintenance patients' ventilation in general anesthesia. It can effectively send narcotic gas into the trachea and allow oxygen ventilation well controlled. However, ETI-related complications such as dental and oral soft tissue injury, intubation and extubation related cardiovascular reactions, hinder its application in some special populations such as elderly patients. Clinical application of laryngeal mask airway (LMA) has brought new options and new ideas for anesthesia management. LMA has the advantage of light damage, small trauma, simple operation and minor cardiovascular response, and it is especially suitable for airway control of patient in short and minimally invasive operation. In recent years, the application of LMA has a greater proportion compared with ETI in some areas. But with LMA application increasing, more and more problems have been reported.

LMA has a greater risk of gastrointestinal reflux and aspiration, because of its inadequate airway tightness. For the same reason, LMA is of intolerance to high airway pressure, and this may lead to hypoventilation in elderly patients with lung compliance or increased airway resistance. At the same time the LMA can't completely prevent incidence of postoperative sore throat and hoarseness. Therefore, it is necessary to carry out a multi-center clinical trial to clarify the peri-operative advantages and disadvantages of LMA to elderly patients, to preliminary explore the LMA complications occurred in elderly patients using predictive models, and to clarify the safety of the LMA in airway support of elderly patients.

1.2 Research Aims The aim of the present research is to study the effects of LMA compared with conventional ETI on elderly patients considering postoperative pulmonary complications, anesthesia and recovery quality, oxygenation and airway support related complications.

1.3 Primary endpoint events Postoperative pulmonary complications before discharge. 1.4 Secondary endpoint events and other pre-specified outcomes 1.4.1 Mortality 1.4.2 PACU stay 1.4.3 Hospiitalization cost and duration 1.4.4 ICU admission and stay time (patients who meet the ICU inclusion criteria are admitted into ICU, those who are admitted into ICU because of bed conversion are excluded, and those who should have been out of ICU are also excluded) 1.4.5 Treatment for PPCs 1.4.6 Blood and sputum culture

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70
* Elective surgery
* BMI ≤ 35 kg/m2
* Provision of signed informed consent

Exclusion Criteria:

* emergency surgery
* have anticipated difficult intubation
* have a broken or unstable cervix
* have laryngeal disease
* are at high risk of aspiration (gastroesophageal reflux disease, full stomach)
* are unable to cooperate for any reason, such as inability to speak or understand, mental disease, or inability to go to the clinics
* have taken experimental drugs in the preceding 3 months or joined another clinical trial
* did not provide informed consent or have withdrawn consent
* are evaluated by the investigator as unsuitable for this trial

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2900 (Actual)
Dates: Start 2016-08-03 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
The occurrence of postoperative pulmonary complications | before discharge
  five-category scale to assess the pulmonary outcomes: 0, no pulmonary complications 1, either one of the following: cough, minor lung atelectasis, dyspnea; 2, cough and sputum, bronchospasm, hypoxemia, atelectasis, hypercapnia; 3, pleural effusion, suspected pneumonia, diagnosed pneumonia, pneumothorax, diagnosed pneumonia, pneumothorax, non-invasive or invasive mechanical ventilation<48hr 4, respiratory failure.

SECONDARY OUTCOMES:
mortality | before discharge
ICU admission rate | before discharge
  Patients who meet the ICU inclusion criteria are admitted into ICU, those who are admitted into ICU because of bed conversion are excluded, and those who should have been out of ICU are also excluded
Hospitalization days | before discharge
PACU stay | before discharge
  PACU stay time collection is based on anesthesia records
Blood and sputum culture | before discharge
  In-hospital medical examinations and tests will be collected
Treatment for PPCs | before discharge
  Included antibiotics, anti-sputum drugs, steroids, mechanical ventilation
ICU stay | before discharge
  Patients who meet the ICU inclusion criteria are admitted into ICU, those who are admitted into ICU because of bed conversion are excluded, and those who should have been out of ICU are also excluded
Hospiitalization cost | before discharge
  Hospitalization cost is collected from hospital bill, regardless of patient's insurerance coverage

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, Ph.D., Study Chair — Department of Anesthesiology Renji Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China

REFERENCES:
- [Background] Patel MG, Swadia V, Bansal G. Prospective randomized comparative study of use of PLMA and ET tube for airway management in children under general anaesthesia. Indian J Anaesth. 2010 Mar;54(2):109-15. doi: 10.4103/0019-5049.63643. PMID 20661347
- [Background] Futier E, Constantin JM, Paugam-Burtz C, Pascal J, Eurin M, Neuschwander A, Marret E, Beaussier M, Gutton C, Lefrant JY, Allaouchiche B, Verzilli D, Leone M, De Jong A, Bazin JE, Pereira B, Jaber S; IMPROVE Study Group. A trial of intraoperative low-tidal-volume ventilation in abdominal surgery. N Engl J Med. 2013 Aug 1;369(5):428-37. doi: 10.1056/NEJMoa1301082. PMID 23902482
- [Background] Wang HE, Szydlo D, Stouffer JA, Lin S, Carlson JN, Vaillancourt C, Sears G, Verbeek RP, Fowler R, Idris AH, Koenig K, Christenson J, Minokadeh A, Brandt J, Rea T; ROC Investigators. Endotracheal intubation versus supraglottic airway insertion in out-of-hospital cardiac arrest. Resuscitation. 2012 Sep;83(9):1061-6. doi: 10.1016/j.resuscitation.2012.05.018. Epub 2012 Jun 1. PMID 22664746
- [Background] Sharma R, Dua CK, Saxena KN. A randomised controlled study comparing the effects of laryngeal mask airway and endotracheal tube on early postoperative pulmonary functions. Singapore Med J. 2011 Dec;52(12):874-8. PMID 22159929
- [Background] Avidan MS, Jacobsohn E, Glick D, Burnside BA, Zhang L, Villafranca A, Karl L, Kamal S, Torres B, O'Connor M, Evers AS, Gradwohl S, Lin N, Palanca BJ, Mashour GA; BAG-RECALL Research Group. Prevention of intraoperative awareness in a high-risk surgical population. N Engl J Med. 2011 Aug 18;365(7):591-600. doi: 10.1056/NEJMoa1100403. PMID 21848460
- [Background] Lerman J, Hammer GB, Verghese S, Ehlers M, Khalil SN, Betts E, Trillo R, Deutsch J; MAPS Investigators Group. Airway responses to desflurane during maintenance of anesthesia and recovery in children with laryngeal mask airways. Paediatr Anaesth. 2010 Jun;20(6):495-505. doi: 10.1111/j.1460-9592.2010.03305.x. Epub 2010 Apr 23. PMID 20456065
- [Background] Ferrari G, Milan A, Groff P, Pagnozzi F, Mazzone M, Molino P, Apra F. Continuous positive airway pressure vs. pressure support ventilation in acute cardiogenic pulmonary edema: a randomized trial. J Emerg Med. 2010 Nov;39(5):676-84. doi: 10.1016/j.jemermed.2009.07.042. Epub 2009 Oct 8. PMID 19818574
- [Background] Zoremba M, Aust H, Eberhart L, Braunecker S, Wulf H. Comparison between intubation and the laryngeal mask airway in moderately obese adults. Acta Anaesthesiol Scand. 2009 Apr;53(4):436-42. doi: 10.1111/j.1399-6576.2008.01882.x. Epub 2009 Feb 18. PMID 19226293
- [Background] Nava S, Hill N. Non-invasive ventilation in acute respiratory failure. Lancet. 2009 Jul 18;374(9685):250-9. doi: 10.1016/S0140-6736(09)60496-7. PMID 19616722
- [Background] Gray AJ, Goodacre S, Newby DE, Masson MA, Sampson F, Dixon S, Crane S, Elliott M, Nicholl J; 3CPO Study Investigators. A multicentre randomised controlled trial of the use of continuous positive airway pressure and non-invasive positive pressure ventilation in the early treatment of patients presenting to the emergency department with severe acute cardiogenic pulmonary oedema: the 3CPO trial. Health Technol Assess. 2009 Jul;13(33):1-106. doi: 10.3310/hta13330. PMID 19615296
- [Background] Glerant JC, Rose D, Oltean V, Dayen C, Mayeux I, Jounieaux V. Noninvasive ventilation using a mouthpiece in patients with chronic obstructive pulmonary disease and acute respiratory failure. Respiration. 2007;74(6):632-9. doi: 10.1159/000105163. Epub 2007 Jul 2. PMID 17622735
- [Background] Severgnini P, Selmo G, Lanza C, Chiesa A, Frigerio A, Bacuzzi A, Dionigi G, Novario R, Gregoretti C, de Abreu MG, Schultz MJ, Jaber S, Futier E, Chiaranda M, Pelosi P. Protective mechanical ventilation during general anesthesia for open abdominal surgery improves postoperative pulmonary function. Anesthesiology. 2013 Jun;118(6):1307-21. doi: 10.1097/ALN.0b013e31829102de. PMID 23542800
- [Background] Biere SS, van Berge Henegouwen MI, Maas KW, Bonavina L, Rosman C, Garcia JR, Gisbertz SS, Klinkenbijl JH, Hollmann MW, de Lange ES, Bonjer HJ, van der Peet DL, Cuesta MA. Minimally invasive versus open oesophagectomy for patients with oesophageal cancer: a multicentre, open-label, randomised controlled trial. Lancet. 2012 May 19;379(9829):1887-92. doi: 10.1016/S0140-6736(12)60516-9. Epub 2012 May 1. PMID 22552194
- [Derived] Zhu L, Shi X, Yin S, Yin J, Zhu Z, Gao X, Jiao Y, Yu W, Yang L. Effectiveness and pulmonary complications of perioperative laryngeal mask airway used in elderly patients (POLMA-EP trial): study protocol for a randomized controlled trial. Trials. 2019 May 8;20(1):260. doi: 10.1186/s13063-019-3351-2. PMID 31068221